CLINICAL TRIAL: NCT04477382
Title: A Prospective, Validation Study to Observe the Effect of House Dust Mite Exposure in an Allergen Exposure Chamber (AEC) Within Dust Mite Allergic Patients Taking an Immune Modulating Dietary Supplement
Brief Title: Impact of a Novel Immune Modulating Dietary Supplement on House Dust Mite Induced Allergic Rhinoconjunctivitis
Status: Completed | Type: Observational
Sponsor: Ecarf Institute GmbH (Other)
Collaborators: Bencard Allergie GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: ImTAEC1
Record Dates: First submitted 2020-07-08; First posted 2020-07-20 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-03

CONDITIONS: Dust Mite Allergy; Allergic Rhinitis
MeSH Terms: conditions — Dust Mite Allergy; Rhinitis, Allergic | interventions — Lactoglobulins; Tretinoin; Zinc

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: holo-BLG (beta-lactoglobulin) - a major component of the protein fraction of raw milk, is loaded with ligands such as retinoic acid, zinc and polyphenol-iron complexes. — Subjects suffering from house dust mite (HDM) allergic rhinoconjunctivitis who are reacting positively to chamber exposure with HDM are reevaluated in the exposure chamber 3 months after taking food supplements.

SUMMARY:
A validated mobile Allergen exposure chamber (AEC) is used to expose qualified study participants suffering from house dust mite (HDM) induced allergic rhinoconjunctivitis. A maximum of four individuals are exposed at a time under standardized conditions with a mixture of allergens from Dermatophagoides pteronyssinus and Dermatophagoides farinae (each 50%, faeces and body allergens; doses of 250 μg/m3 air; 21°C, and 55% relative air moisture). After the first exposure, a dietary supplement lozenge, containing beta-lactoglobulin (BLG), iron, retinoic acid, zinc and polyphenols, is taken twice daily for a period of 12 weeks, followed by the second exposure. A minimum of thirty persons are challenged with HDM allergen. After entering the chamber there is an acclimatization phase of 20 minutes with no exposure. Exposure time starts after acclimatization in the chamber and is 120 minutes at each visit. Objective parameters are recorded every 30 minutes, and subjective parameters are recorded every 10 minutes over a period of 120 minutes. During the exposure a plateau (steady-state) of total nasal symptom score with a difference from baseline is measured in all participants for each of the two exposures with HDM.

ELIGIBILITY:
Inclusion Criteria:

* Allergy to house dust mite (HDM) with rhinoconjunctivitis symptoms with/without asthma. These allergic symptoms must have been present for at least 2 years and severity assessed by anamnesis according to ARIA guidelines (mild; moderate/severe - Bousquet et al, 2007)
* Positive skin test to HDM extract using a skin testing diagnostic product used in the daily routines of the clinics, with a wheal diameter > 3 mm
* Positive nasal provocation test to HDM allergen as used in the chamber and/or a history of TNSS ≥ 3 after 120 min HDM exposure in the chamber
* Oral and written informed consent

Exclusion Criteria:

* Current or previous treatment with allergy vaccination within the last two years.
* Concomitant (or newly developing during study period) severe disease interfering with allergy testing
* Co-medication interfering with allergy testing for other diseases, e.g. immunosuppressants, oral and/or nasal corticosteroids, chromones and pregnancy
* Clinically relevant co-sensitization to early blossoming tree pollen allergens, and cat allergens
* Patient with FEV1 < 80% of predicted value prior to exposure
* Patients with severe asthma and / or with a history of uncontrolled asthmatic attacks in the last three months before the selection process
* Patients with an upper intestinal tract disease, where the local examiner believes that taking the dietary supplement could pose a risk to the patient
* History of serious chronic medical conditions and/or any disease where, in the opinion of the site investigator, participation in the trial would pose a risk for the patient
* Treatment prior to study visits and during the whole study time with:

  * systemic corticosteroids within three weeks (21 days)
  * topical nasal corticosteroids within two weeks (14 days)
  * chromones within 7 days
  * antihistamines within 72 hours before visit 1
  * antibiotics within 3 months before visit 1 and during the whole study
  * anti-allergic drugs during the whole study time.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study group recruitment is based on an existing data base of subjects suffering from HDM-induced allergic rhinoconjunctivitis reacting positively to chamber exposure with HDM and by advertising for volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
TNSS | After 120 minutes of allergen challenge
  Total Nasal Symptom Score (TNSS) in response to HDM exposure in an AEC at V1 (baseline AEC exposure) versus V3 (final AEC exposure). The TNSS is the sum of 4 nose symptoms (runny nose, sneezing, itchy nose, and blocked nose) on a scale of 0 to 3 (no symptoms, mild symptoms, moderate symptoms, and severe symptoms), leading to a maximum TNSS of 12.

SECONDARY OUTCOMES:
TSS | Up to 120 minutes following allergen challenge
  Total Symptom Score in response to HDM exposure in an AEC at V1 (baseline AEC exposure) versus V3 (final AEC exposure). The TSS is the sum of 4 nose symptoms (runny nose, sneezing, itchy nose, and blocked nose), 3 eye symptoms (itchy eyes, watery eyes, and gritty feeling), 4 bronchial symptoms (wheezing, cough, breathlessness, and asthma), and 2 other symptoms (itchy palate, and itchy skin) on a scale of 0 to 3 (no symptoms, mild symptoms, moderate symptoms, and severe symptoms), leading to a maximum TSS of 39.
TESS | Up to 120 minutes following allergen challenge
  The Total Eye Symptom Score (TESS) is the sum of 3 eye symptoms (itchy eyes, watery eyes, and gritty feeling) on a scale of 0 to 3 (no symptoms, mild symptoms, moderate symptoms, and severe symptoms), leading to a maximum TESS of 9.
TBSS | Up to 120 minutes following allergen challenge
  The Total Bronchial Symptom Score (TBSS) is the sum of 4 bronchial symptoms (wheezing, cough, breathlessness, and asthma) on a scale of 0 to 3 (no symptoms, mild symptoms, moderate symptoms, and severe symptoms), leading to a maximum TBSS of 12.
VAS | Recorded at time zero (0) and every 30 minutes during exposure until 120 minutes
  Visual Analogue Scale: Before, every 30 minutes during and after the exposure patients grade the question on their well-being by putting a vertical line on a 10 cm line representing severity from 0 cm "very good" to 10 cm "very bad".
PNIF | Recorded at time zero (0), and every 30 minutes during exposure until 120 minutes. An acclimatization phase of 20 minutes takes place in the chamber - so time point zero is when exposure starts after 20 minutes of acclimatization
  PNIF (peak nasal inspiration flow) liter/minute.
PEF | Recorded at time zero (0) and every 30 minutes during exposure until 120 minutes. An acclimatization phase of 20 minutes takes place in the chamber - so time point zero is when exposure starts after 20 minutes of acclimatization
  PEF (peak expiratory flow) liter/minute.
FEV1 | Up to 120 minutes following allergen challenge
  Forced expiratory volume in 1 second, before and after the exposure.
FEV1/FVC | Up to 120 minutes following allergen challenge
  Forced expiratory volume in 1 second/forced vital capacity ratio, before and after the exposure.
Need for rescue medication and/or emergency treatment | up to 24 hours after AEC exposure
  Need for rescue medication and/or emergency treatment.
Adverse events with regard to the taken dietary supplement | up to 24 hours after the final AEC exposure
  Number of events and number of patients recording adverse events with regard to the taken dietary supplement. After completing the baseline AEC exposure at V1 the patients will enter the 3-month consumption period with the dietary supplement. Every patient will document potential AEs in the patient report form. In addition, the patient will be called every 4 weeks during the consumption period to follow up on potential AEs with the intake. The final safety phone call will be made 24 hours after the final AEC exposure.
Adverse events with regards to the allergen exposure | up to 24 hours after AEC exposure
  Number of events and number of patients recording late-phase reactions and/or adverse events with regards to the allergen exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Becker, Study Director — Managing Director, ECARF Institute GmbH
Locations (1):
- ECARF Institute GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bergmann KC, Graessel A, Raab J, Banghard W, Krause L, Becker S, Kugler S, Zuberbier T, Ott V, Kramer MF, Roth-Walter F, Jensen-Jarolim E and Guethoff S. Targeted micronutrition via holo-BLG based on the farm effect in house dust mite allergic rhinoconjunctivitis patients - first evaluation in a standardized allergen exposure chamber. Allergo Journal International. 2021. doi:10.1007/s40629-021-00163-9.